CLINICAL TRIAL: NCT06148974
Title: Effects of Oat and Oat Components on Cardiometabolic- and Cognitive Test Variables
Brief Title: Effects of Plant Polar Lipids on Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Nilsson (Other)
Responsible Party: Sponsor-Investigator, Anne Nilsson, Associate professor, Lund University
Organization: Lund University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Prot.2018/8-23
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Due to the character of the test products, the masking is partial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Polar lipid 1 (Experimental): 15 g Plant polar lip 1 consumed with a white wheat bread including 50 g available carbohydrates
  Interventions: Dietary Supplement: Polar lipid 1
- Polar lipid 2 (Experimental): 15 g Plant polar lipids 2 consumed with a white wheat bread including 50 g available carbohydrates
  Interventions: Dietary Supplement: Polar lipid 2
- non-polar lipids (Active Comparator): 15 g commonly consumed non-polar lipids consumed with a white wheat bread including 50 g available carbohydrates
  Interventions: Dietary Supplement: Non-polar lipids
- no lipids (Placebo Comparator): A white wheat bread including 50 g available carbohydrates
  Interventions: Other: No lipids

INTERVENTIONS:
Dietary Supplement: Polar lipid 1 — 15g plant polar lipids from plant source 1. The lipid supplement is consumed spread on a commercial white wheat flour bread as a source of available carbohydrates (50 g).
  Arms: Polar lipid 1
Dietary Supplement: Polar lipid 2 — 15g plant polar lipids from plant source 2. The lipid supplement is consumed spread on a commercial white wheat flour bread as a source of available carbohydrates (50 g).
  Arms: Polar lipid 2
Dietary Supplement: Non-polar lipids — 15g non-polar plant lipids from plant source 1. The lipids supplement is consumed spread on a commercial white wheat flour bread as a source of available carbohydrates (50 g).
  Arms: non-polar lipids
Other: No lipids — A commercial white wheat flour bread as a source of available carbohydrates (50 g), without added lipids.
  Arms: no lipids

SUMMARY:
In this randomized controlled trial, two different plant polar lipids are investigated with respect to their potential to affect acute and second meal glucose tolerance and appetite sensations. The effects are compared with a common non-polar commercial oil. The lipids are consumed spread on a white wheat bread. A white wheat bread without added lipids is included as a control product. The test products are consumed at breakfast, and test variables are investigated in the postprandial period after the test breakfast and also after a second meal standard lunch.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women
* non-smokers
* between 20-40 years of age
* BMI between 18,5-30 kg/m2
* No known metabolic disorders or food allergies.
* The test subjects should follow a normal diet in accordance with the Nordic Nutrition Recommendations.

Exclusion Criteria:

* Fasting blood glucose ≥6.1 mmol/L
* Use of antibiotics or probiotics in the last three months or during the study period.
* Smoking
* Blood donation during the last two months and during the study.
* Food allergies or food intolerances
* Cardiovascular diseases
* Metabolic diseases
* Inflammatory bowel diseases.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentration (glucose tolerance) | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Blood glucose will be determined repeatedly after the breakfast and also following a standardised lunch. The primary outcome measures for glucose concentrations are incremental areas under the curve after the test breakfast and after the standardised lunch

SECONDARY OUTCOMES:
Serum insulin concentrations | 5.5 hours. Fasting (time =0), 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Insulin will be determined repeatedly after the breakfast and also following a standardised lunch. The primary outcome measures for insulin are incremental areas under the curve after the test breakfast and after the standardised lunch
Subjective hunger sensations | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Subjective appetite variables will be determined repeatedly after the breakfast and also following a standardised lunch. The secondary outcome measures are areas under the curve after the test breakfast and after the standardised lunch. Subjective appetite variables will be determined using a 100 mm Visual Analogue Scale (VAS).
Subjective satiety sensations | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Subjective appetite variables will be determined repeatedly after the breakfast and also following a standardised lunch. The secondary outcome measures are areas under the curve after the test breakfast and after the standardised lunch. Subjective appetite variables will be determined using a 100 mm Visual Analogue Scale (VAS).
Subjective sensations of desire to eat | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Subjective appetite variables will be determined repeatedly after the breakfast and also following a standardised lunch. The secondary outcome measures are areas under the curve after the test breakfast and after the standardised lunch. Subjective appetite variables will be determined using a 100 mm Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, dep of Food Technology, Engineering, and Nutrition, Lund, Välj..., Sweden

IPD SHARING:
Plan to Share IPD: No